CLINICAL TRIAL: NCT06891222
Title: Integrating Electrocardiogram and Focused Cardiac Ultrasound for Enhanced Cardiac Disease Screening; Structural Cardiac Assessment With Networked AI-ECG & FOCUS (SCAN) Study
Brief Title: A Study of Electrocardiogram and Focused Cardiac Ultrasound for Enhanced Cardiac Disease Screening
Acronym: SCAN
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Gal Tsaban, Principal Investigator, Mayo Clinic
Other Study IDs: 25-000609
Record Dates: First submitted 2025-03-18; First posted 2025-03-24 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Cardiac Disease
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Integrated pathway
  Interventions: Diagnostic Test: AI-ECG (artificial intelligence-enabled electrocardiogram); Diagnostic Test: Focus Screening (focused cardiac ultrasonography)
- Standard of Care pathway

INTERVENTIONS:
Diagnostic Test: AI-ECG (artificial intelligence-enabled electrocardiogram) — Participants will undergo electrocardiogram analysis using AI-ECG during the baseline visit
  Groups: Integrated pathway
Diagnostic Test: Focus Screening (focused cardiac ultrasonography) — Participants will undergo a focused cardiac ultrasound if the AI-ECG reflects a positive value
  Groups: Integrated pathway

SUMMARY:
The purpose of this study is to evaluate and compare the effectiveness of active screening for SHD in asymptomatic outpatients referred for an ECG, using a combination of AI-ECG and FOCUS. Invites will be sent and participants enrolled electronically.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years of age)
* Echocardiogram is not clinically indicated

Exclusion Criteria:

* Prior history of congenital or acquired SHD, as defined by the following

  1. Aortic Stenosis:
  2. Heart Failure
  3. Left Ventricular Dysfunction
  4. Cardiac Amyloidosis
  5. Hypertrophic Cardiomyopathy (HCM)
  6. Rheumatic Heart Disease
  7. Congenital Heart Disease
* Recent (within last 12 months) echocardiogram
* Scheduled clinically indicated future echocardiogram
* Inability to provide informed consent to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All subjects aged 18 or older without known congenital or acquired SHD scheduled to undergo an elective outpatient electrocardiogram
Sampling Method: Probability Sample
Enrollment: 10500 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects to be diagnosed with SHD (structural heart disease) | Baseline, 6 months, 1 year
  Percentage of subjects to be diagnosed with SHD will be determined by the number of subjects that have a positive SHD screening. Positive SHD screening is defined by any one of the following: decreased LVEF (left ventricular ejection fraction), cardiac amyloidosis, aortic stenosis, and hypertrophic cardiomyopathy.
Positive predictive value (PPV) | Baseline, 6 months, 1 year
  Positive predictive value (PPV) will be measured as a percentage. PPV will reflect the percentage of times that each screening pathway matches a formal echocardiogram diagnosis.

SECONDARY OUTCOMES:
Number of deaths | 1 year
  Number of deaths will include all-cause deaths.
Number of adverse cardiovascular events | 1 year
  Number of adverse cardiovascular events includes systolic heart failure, rt failure hospitalization.
Percentage of subjects to be diagnosed with decreased LVEF (left ventricular ejection fraction) | Baseline, 6 months,1 year
  Percentage of subjects to be diagnosed with decreased LVEF will be determined by the percentage of subjects to have a LVEF lower than 50%.
Percentage of subjects to be diagnosed with cardiac amyloidosis | Baseline, 6 months,1 year
  Percentage of subjects to be diagnosed with cardiac amyloidosis will be determined by the number of subjects that have a positive AI-ECG or ultrasound. Cardiac amyloidosis is the buildup of protein in the heart muscle that affect the structure and function of the heart.
Percentage of subjects to be diagnosed with aortic stenosis | Baseline, 6 months,1 year
  Percentage of subjects to be diagnosed with aortic stenosis will be determined by the number of subjects that have a positive AI-ECG or ultrasound. Aortic stenosis is the narrowing of the aortic value decreasing the blood flow from heart to the aorta.
Percentage of subjects to be diagnosed with hypertrophic cardiomyopathy | Baseline, 6 months,1 year
  Percentage of subjects to be diagnosed with hypertrophic cardiomyopathy will be determined by the number of subjects that have a positive AI-ECG or ultrasound. Hypertrophic cardiomyopathy is the thickening of the heart muscle which leads to reduced blood flow.

CONTACTS AND LOCATIONS:
Overall Officials: Gal Tsaban, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No